CLINICAL TRIAL: NCT06551142
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of GSK5764227 as Monotherapy and in Combination in Participants With Advanced Solid Tumors
Brief Title: A Study of GSK5764227 in Participants With. Advanced Solid Tumors (EMBOLD PanTumor-101)
Acronym: PanTumor-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 223054; 2024-513663-10 (EudraCT Number)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms
Keywords: Solid Tumors; GSK5764227; Neoplasms; EMBOLD PanTumor-101
MeSH Terms: conditions — Neoplasms | interventions — Cisplatin; Carboplatin; atezolizumab; pembrolizumab; durvalumab; Cetuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1a: Dose escalation-GSK5764227 Monotherapy (Experimental)
  Interventions: Biological: GSK5764227
- Phase 1a- Dose escalation- Combination therapy (Experimental)
  Interventions: Biological: GSK5764227; Drug: Cisplatin; Drug: Carboplatin; Biological: Atezolizumab; Biological: Pembrolizumab; Biological: Durvalumab; Biological: Cetuximab; Biological: Bevacizumab
- Phase 1b- Dose optimisation/ expansion (Experimental)
  Interventions: Biological: GSK5764227; Biological: Atezolizumab

INTERVENTIONS:
Biological: GSK5764227 — GSK5764227 will be administered
Drug: Cisplatin — Cisplatin will be administered
  Arms: Phase 1a- Dose escalation- Combination therapy
Drug: Carboplatin — Carboplatin will be administered
  Arms: Phase 1a- Dose escalation- Combination therapy
Biological: Atezolizumab — Atezolizumab will be administered
  Arms: Phase 1a- Dose escalation- Combination therapy; Phase 1b- Dose optimisation/ expansion
Biological: Pembrolizumab — Pembrolizumab will be administered
  Arms: Phase 1a- Dose escalation- Combination therapy
Biological: Durvalumab — Durvalumab will be administered
  Arms: Phase 1a- Dose escalation- Combination therapy
Biological: Cetuximab — Cetuximab will be administered
  Arms: Phase 1a- Dose escalation- Combination therapy
Biological: Bevacizumab — Bevacizumab will be administered
  Arms: Phase 1a- Dose escalation- Combination therapy

SUMMARY:
The goal of this study is to assess the safety, tolerability, clinical activity and pharmacokinetics of GSK5764227. The study will also see how the levels of GSK5764227 will change over time at different dose amounts when administered alone and in combination with other medicines like carboplatin, cisplatin, atezolizumab, pembrolizumab, durvalumab, bevacizumab, cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants at least 18 years of age (≥18 years)
* Participants with histologically confirmed advanced/metastatic solid tumors, as defined per study phase and cohort, as follows:

  o Phase 1a:
  * Participants with advanced/metastatic solid tumors.
  * For monotherapy dose escalation: participants must have progressed on or become intolerant to all available SOC therapies.
  * For combination dose escalation: participants must have received 3 or fewer prior lines of systemic anticancer therapy in the advanced/metastatic setting
* Has at least 1 target lesion per RECIST 1.1, as determined by the investigator.
* Has an ECOG performance status of 0 or 1, with no deterioration in the 2 weeks before first dose.
* Has adequate organ function.
* Where available, participants should provide a formalin fixed and paraffin embedded (FFPE) tumor sample from the most recent biopsy of primary cancer or from a metastatic site for central testing. Tumor tissue is necessary for retrospective detection of B7 homolog 3 protein (B7-H3) expression by Immunohistochemistry (IHC) and other biomarker analysis.
* At least one of the following treatment combinations/monotherapy (a, b, c, or d) is clinically indicated:

  1. Atezolizumab, durvalumab, or pembrolizumab in combination with cisplatin or carboplatin (for combination 1 only).
  2. Atezolizumab, durvalumab, or pembrolizumab as monotherapy (for combination 2 only)
  3. Bevacizumab as monotherapy (for combination 3 only)
  4. Cetuximab as monotherapy (for combination 4 only)
* Additional inclusion criteria for Phase 1b Chinese participants:

Chinese participants are considered eligible if they meet all of the following:

* Born in mainland China, Hong Kong or Taiwan
* Descendant of 2 ethnic Chinese parents and 4 ethnic Chinese grandparents
* All participants who do not meet either of the above-mentioned inclusion criteria for Chinese participants will be considered as global (non-Chinese) participants.

Exclusion Criteria:

* Has ongoing adverse reaction(s) from prior therapy that has(have) not recovered to ≤Grade 1 or to the baseline status preceding prior therapy.
* Prior treatment with orlotamab, enoblituzumab, I-Dxd, or other B7-H3 targeted agents.
* Primary brain tumor or evidence of brain metastasis (unless meeting the following criteria at the same time: asymptomatic; medically stable for at least 4 weeks prior to initial dosing; no steroid treatment required for at least 4 weeks prior to initial dosing; and no midline shift due to herniation); or untreated progression due to brain metastasis or primary brain tumor during or after the last treatment prior to screening; or evidence of meningeal/brainstem involvement; or evidence of spinal cord compression (detected by radiographic examination, symptomatic or not).
* Any of the following cardiac examination abnormality:

  * Has QT interval, corrected for heart rate (QTc) >450 msec or QTc >480 msec for participants with bundle branch block.
  * Evidence of current clinically significant arrhythmias or ECG abnormalities (e.g., complete left bundle branch block, third-degree atrioventricular [AV] block, second-degree AV block, PR interval >250 msec).
  * Risk factors of prolonged QTc or arrhythmia events, such as heart failure, refractory hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death of any direct relative under 40 years old or any concomitant medications that prolong the QT interval.
  * Left ventricular ejection fraction (LVEF) <50%.
* Has severe, uncontrolled or active CV disorders, serious or poorly controlled hypertension, clinically significant bleeding symptoms or serious arteriovenous thromboembolic events Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids.
* Has donated blood or blood products in excess of 500 mL (approximately 1 pint) within one month prior to first dose of study treatment.
* Has a history of autoimmune disease that has required systemic treatments in the 2 years prior to screening. Participants with prior history of autoimmune disease must be discussed with the medical monitor. Replacement therapy is not considered a form of systemic therapy (e.g., thyroid hormone for autoimmune thyroiditis or insulin is not exclusionary).
* Has any history of prior allogenic or autologous bone marrow transplant or other solid organ transplant.
* Has received immunosuppressive agents within 30 days prior to first dose of study treatment (or requires long-term (30 days or longer) glucocorticoid therapy). Low-dose corticosteroids (prednisone ≤10 mg/day or equivalent) may be administered. Use of inhaled or topical steroids and prophylactic corticosteroids for procedures are permitted.
* Participants in dehydrated condition.
* Participant with history of nephrotic syndrome or Grade 3 proteinuria. Participants discovered to have ≥2 proteinuria on dipstick at screening should undergo a 24-hour urine collection and must demonstrate <2 g of protein in 24 hours to be eligible.
* History of abdominal or gastrointestinal fistula, tracheoesophageal fistula or any Grade 4 fistula, gastrointestinal perforation, intra-abdominal abscess or active clinical concern for bowel obstruction.
* Has any active renal condition (e.g., requirement for dialysis, or any other significant renal condition that could affect the participant's safety). NOTE: renal obstruction successfully managed by stenting is permitted.

Additional exclusion criteria for participants receiving combination therapy

* Has received prior systemic anticancer therapy within 28 days of first dose of study treatment (combinations 1, 3 and 4 only).
* Has experienced any of the following with prior immunotherapy: any immune-mediated adverse event [imAE] ≥ Grade 3, immune-mediated severe neurologic events of any-grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain-Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade (Stevens-Johnson syndrome [SJS], Toxic epidermal necrolysis [TEN], or Drug reaction with eosinophilia and systemic symptoms [DRESS] syndrome), symptomatic pericarditis of any etiology within 6 months prior to the administration of study intervention, or myocarditis of any grade. Clinically significant laboratory abnormalities, as judged by investigator, are not exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-09-24 (Estimated); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of participants with Adverse Events (AEs) | Up to approximately 28 months
Phase 1a: Number of participants with Dose Limiting Toxicities (DLTs) | Up to 21 days
Phase 1a: Number of participants with AEs, serious adverse events (SAEs) and adverse events of special interest (AESIs) by severity | Up to approximately 30 months
Phase 1a: Number of participants with AEs leading to dose modifications | Up to approximately 28 months
Phase 1a: Number of participants with changes in vital signs, body weight, laboratory tests, electrocardiogram (ECG) and Eastern Cooperative Oncology Group (ECOG) performance status | Up to approximately 28 months
Phase 1b: Confirmed Objective Response Rate (cORR) | Up to approximately 27 months
  cORR is defined as the proportion of participants who have confirmed Complete response (CR) or Partial response (PR), assessed by the investigator according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST V1.1) criteria or other imaging criteria for defined tumor types.

SECONDARY OUTCOMES:
Phase 1a and Phase 1b: Maximum concentration (Cmax) of GSK5764227 | Up to approximately 28 months
Phase 1a and Phase 1b: Time to reach maximum concentration (Tmax) of GSK5764227 | Up to approximately 28 months
Phase 1a and Phase 1b: Area under the curve (AUC) of GSK5764227 | Up to approximately 28 months
Phase 1a and Phase 1b: Trough concentration (Ctrough) of GSK5764227 (conjugated antibody) | Up to approximately 28 months
Phase 1a and Phase 1b: Trough concentration (Ctrough) of GSK5764227 (total antibody) | Up to approximately 28 months
Phase 1a and Phase 1b: Trough concentration (Ctrough) of GSK5757810 (small-molecule toxin) | Up to approximately 28 months
Phase 1a: Confirmed Objective Response Rate (cORR) | Up to approximately 33 months
  cORR is defined as the proportion of participants who have confirmed CR or PR, per RECIST V1.1 by investigator
Phase 1a: Disease control rate at 12 weeks (DCR12) | At 12 weeks
  DCR is defined as the proportion of participants who have achieved CR, PR or Stable disease (SD) ≥11 weeks per RECIST v1.1 by investigator assessment
Phase 1b: Disease control rate at 12 weeks (DCR12) | At 12 weeks
  DCR defined as the proportion of participants who have achieved CR, PR or SD ≥11 weeks per RECIST 1.1 or other imaging criteria for defined tumor types by investigator.
Phase 1a: Duration of Response (DoR) | Up to approximately 33 months
  DoR is defined as the date of first documented objective response (CR/PR) until per RECIST 1.1 by investigator assessment to the date of first documented PD or death due to any cause, whichever comes first.
Phase 1b: Duration of Response (DoR) | Up to approximately 33 months
  DoR defined as the time from the date of first documented objective response (CR/PR) per RECIST 1.1 or other imaging criteria for defined tumor types by investigator assessment to the date of first documented PD or death due to any cause, whichever comes first.
Phase 1b: Proportion of Participants with Tumour antigen Decrease From Baseline >=50% response rate | Up to approximately 33 months
  Tumour antigen response rate is defined as a proportion of participants with ≥50% decrease from baseline in the tumour antigen during the study. Any observed ≥50% decrease will be confirmed by repeat assessment after approximately 3 weeks
Phase 1a and Phase 1b: Number of participants with Antidrug antibody (ADA) or Neutralizing Antibody (NAb) | Up to approximately 30 months
Phase 1a and Phase 1b: Titers of ADA against GSK5764227 | Up to approximately 30 months
Phase 1b: Number of participants with AEs, SAEs and AESI by severity | Up to approximately 30 months
Phase 1b: Number of participants with AEs leading to dose modifications | Up to approximately 27 months
Phase 1b: Number of participants with changes in vital signs, body weight, laboratory tests, ECG, ECHO and ECOG performance status | Up to approximately 28 months
Phase 1b: Progression-Free Survival (PFS) | Up to approximately 33 months
  PFS is defined as the time from the date of first dose (dose expansion) or date of randomization (dose optimization) until the earliest date of documented disease progression (investigator-assessed according to RECIST 1.1 or other imaging criteria for defined tumor types) or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (14):
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Myrtle Beach, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, West Valley City, Utah
  - GSK Investigational Site, Norfolk, Virginia
- Argentina (2):
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Viedma
- Canada (4):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- France (3):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Villejuif
- Italy (2):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
- Japan (4):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Panama City, Panama
- South Korea (2):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
- Taiwan (5):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- United Kingdom (4):
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/